CLINICAL TRIAL: NCT01023087
Title: The Incidence of Renal Impairment Associated With Polymyxin E Treatment and the Impact of Measuring Colistin Levels
Brief Title: Renal Impairment Associated With Colistin Levels
Status: Completed | Type: Observational
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Dr. Moshe Hersch, Shaare Zedek Medical Center, Jerusalem, Israel
Other Study IDs: COLISTIN.RF.10
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2010-07

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Colistin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Separated blood samples for Colistin levels assesment are kept in the immunology department refrigirator for analysis when the immunological method of the blood Colistin levels will be ready for use.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treatment: Patients with sepsis treated with polymyxin E (colistin)
  Interventions: Drug: Polymyxin E (Colistin)
- Control: Patients with sepsis treated with other, non-nephrotoxic antibiotic medication
  Interventions: Drug: Non-nephrotoxic antibiotics

INTERVENTIONS:
Drug: Polymyxin E (Colistin) — Antibiotic medication; dosage to be decided according to infectious disease consultant recommendation.
  Other Names: Coliracin
  Groups: Treatment
Drug: Non-nephrotoxic antibiotics — To be decided by the infectious disease consultant
  Other Names: Non-nephrotoxic antibiotics, as required
  Groups: Control

SUMMARY:
Colistin is a relatively old antibiotic drug which its use has been abandoned through the 1970s because it was considered nephrotoxic.

Recently ( the last decade) it has been reappraised because multidrug resistant Gram negative bacteria have emerged causing life threatening infections with no other good enough treatment. Moreover, more controlled studies from the recent years show less toxic effect of the drug.

The investigators' study is a prospective study comparing renal function in a group of hospitalized patients with sepsis (infection) receiving intravenous treatment with Colistin (antibiotics) with a control group which its patients receive other non nephrotoxic antibiotics.

The investigators' study hypothesis is that patients receiving Colistin would have renal function decline in higher rates than those seen usually in hospitalized patients in the Internal medicine wards with sepsis.

Another goal of the study is to find correlation between Colistin levels in the plasma (after Colistin reaches steady state) and nephrotoxicity seen during or after use of this drug.

DETAILED DESCRIPTION:
Colistin is a relatively old antibiotic drug which its use has been abandoned through the 1970s because it was considered nephrotoxic.

Recently ( the last decade) it has been reappraised because multidrug resistant Gram negative bacteria have emerged causing life threatening infections with no other good enough treatment. Moreover, more controlled studies from the recent years show less toxic effect of the drug.

The investigators' study is a prospective study comparing renal function in a group of hospitalized patients with sepsis (infection) receiving intravenous treatment with Colistin (antibiotics) with a control group which its patients receive other non nephrotoxic antibiotics.

The investigators' study hypothesis is that patients receiving Colistin would have renal function decline in higher rates than those seen usually in hospitalized patients in the Internal medicine wards with sepsis.

Another goal of the study is to find correlation between Colistin levels in the plasma (after Colistin reaches steady state) and nephrotoxicity seen during or after use of this drug.The measurement of the Colistin levels are planned to be done by immunological methods, by developing specific antibodies to Colistin in a laboratory in France.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients diagnosed with sepsis requiring antibiotic treatment
* Age 18 years old and above
* Gender - male or female

Exclusion Criteria:

* Anticipated antibiotic treatment of less than 7 consecutive days
* Concurrent treatment with other nephrotoxic antibiotic drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the Department of Internal Medicine with sepsis of any origin.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2009-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Serum creatinine changes. | Blood examination every 3 days until discharge

SECONDARY OUTCOMES:
Mortality | During hospitalization
Correlation between creatinine levels and colistin levels | During hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Hersch, MD; MSc., Study Chair — Shaare Zedek Medical Center, Jerusalem
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel